CLINICAL TRIAL: NCT01816906
Title: Development of a New Generation of DIABetic Footwear Using an Integrated Approach and SMART Materials
Brief Title: Development and Testing of a New Generation of Diabetic Footwear
Acronym: DiaBSmart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Staffordshire University (Other)
Collaborators: India Diabetes Research Foundation & Dr. A. Ramachandran's Diabetes Hospitals (Other)
Responsible Party: Principal Investigator, Nachiappan Chockalingam, Director, Biomechanics Facility, Staffordshire University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DiaBSmart-01; DiaBSmart -2011-IAPP (Other Grant/Funding Number: FP7-PEOPLE-2011-IAPP Grant Agreement Number 285985)
Record Dates: First submitted 2013-03-14; First posted 2013-03-22 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Complications; Diabetic Neuropathies
MeSH Terms: conditions — Diabetes Complications; Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCP Insole (Active Comparator): The intervention is "Footwear: MCP". MCP insoles are commonly used within Diabetic sandals in India.
  Interventions: Device: Footwear: MCP
- PU insole (Active Comparator): The intervention is "Footwear: PU". Insoles made of Polyurethane(PU) are given to the participants in the intervention arm.
  Interventions: Device: Footwear :PU

INTERVENTIONS:
Device: Footwear :PU — One group of patients will receive "Footwear" with PU insoles
  Arms: PU insole
Device: Footwear: MCP — One group of patients will receive footwear with MCP insoles
  Arms: MCP Insole

SUMMARY:
This particular trial is looking to compare the effectiveness of two types of foot bed/ sole materials used within diabetic footwear.

DETAILED DESCRIPTION:
DiaBSmart as a project aims to generate, transfer and exchange the clinical, academic and production knowledge between the partners to create a new generation of diabetic footwear through a newly developed patient assessment system. The transfer of knowledge between various sectors ensures that the need of patients is considered and transferred effectively to product development using a scientific approach. The objectives include:(1) the design and development of an integrated system of DIABetic foot assessment (2) to validate the newly developed system using experimental methods (3) to develop a suitable material to meet the mechanical and clinical requirements (4) to evaluate the mechanical and clinical effectiveness of material choice in reducing the potential risk of foot complications. The Numerical, Experimental and Mathematical Analyses system will integrate all aspects of diabetic footwear including; clinical and biomechanical assessment, material choice and aesthetic design. Proposed interdisciplinary, inter-sectorial approach is unique and brings together the expertise from research institutions, industry and clinics. This project while enhancing the knowledge base in diabetic assessment; will have a clear impact on new product development leading to both clinical and economic benefits. The products include a new generation of integrated SMART /multi material midsoles and/or orthoses for diabetic footwear. Properties of the materials will be optimised with a view to minimise/ redistribute the pressure and hence the stress on the soft tissue in the critical plantar areas of the foot. Whilst significantly affecting the course of the disease, the products will aim to reduce the risk of limb loss in patients with diabetes, the most frequent cause of non-traumatic lower-limb amputations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Diabetes by WHO criteria
* Lack of sensation to 10 g monofilament or VPT >25 V
* Ability to walk independently for 10 m
* No ambulatory status
* No severe foot deformity like Charcot foot
* Willingness to be assigned to randomisation of footwear
* At least one palpable pedal pulse on each foot

Exclusion Criteria:

* Previous ulceration or current Trophic Ulcers
* Active foot infection
* Alzheimer and dementia and impaired cognitive function
* Gross abnormality or Foot deformity requiring footbed customisation
* Chronic Kidney Disease
* Hammer toes
* Previous foot surgeries

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nachiappan Chockalingam, PhD, Principal Investigator — Staffordshire University; Lakshmi Sundar, MBBS, Study Director — AR Hospitals/ IDRF; Roozbeh Naemi, PhD, Study Director — Staffordshire University
Locations (1):
- IDRF/ AR Hopsitals, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatzistergos PE, Naemi R, Chockalingam N. An MRI compatible loading device for the reconstruction of clinically relevant plantar pressure distributions and loading scenarios of the forefoot. Med Eng Phys. 2014 Sep;36(9):1205-11. doi: 10.1016/j.medengphy.2014.06.006. Epub 2014 Jul 7. PMID 25012640
- [Background] Naemi R, Chatzistergos PE, Chockalingam N. A mathematical method for quantifying in vivo mechanical behaviour of heel pad under dynamic load. Med Biol Eng Comput. 2016 Mar;54(2-3):341-50. doi: 10.1007/s11517-015-1316-5. Epub 2015 Jun 5. PMID 26044551
- [Background] Healy A, Naemi R, Chockalingam N. The effectiveness of footwear and other removable off-loading devices in the treatment of diabetic foot ulcers: a systematic review. Curr Diabetes Rev. 2014;10(4):215-30. doi: 10.2174/1573399810666140918121438. PMID 25245020
- [Background] Healy A, Naemi R, Chockalingam N. The effectiveness of footwear as an intervention to prevent or to reduce biomechanical risk factors associated with diabetic foot ulceration: a systematic review. J Diabetes Complications. 2013 Jul-Aug;27(4):391-400. doi: 10.1016/j.jdiacomp.2013.03.001. Epub 2013 May 1. PMID 23643441
- [Background] NAEMI, R., HEALY, A., Sundar, L., Ramachandran, A.R. and CHOCKALINGAM, N., 2013. A Combined Technique for Randomisation of a Small Number of Participants with a Variety of Covariates into Treatment and Control Groups in Randomised Controlled Trials. Journal of Clinical Trials, 4(01).
- [Result] Chatzistergos PE, Naemi R, Healy A, Gerth P, Chockalingam N. Subject Specific Optimisation of the Stiffness of Footwear Material for Maximum Plantar Pressure Reduction. Ann Biomed Eng. 2017 Aug;45(8):1929-1940. doi: 10.1007/s10439-017-1826-4. Epub 2017 May 9. PMID 28484892
- [Result] Healy A, Naemi R, Sundar L, Chatzistergos P, Ramachandran A, Chockalingam N. Hallux plantar flexor strength in people with diabetic neuropathy: Validation of a simple clinical test. Diabetes Res Clin Pract. 2018 Oct;144:1-9. doi: 10.1016/j.diabres.2018.07.038. Epub 2018 Aug 13. PMID 30114460
- [Result] Naemi R, Chatzistergos P, Suresh S, Sundar L, Chockalingam N, Ramachandran A. Can plantar soft tissue mechanics enhance prognosis of diabetic foot ulcer? Diabetes Res Clin Pract. 2017 Apr;126:182-191. doi: 10.1016/j.diabres.2017.02.002. Epub 2017 Feb 10. PMID 28259007
- [Result] Naemi R, Chatzistergos P, Sundar L, Chockalingam N, Ramachandran A. Differences in the mechanical characteristics of plantar soft tissue between ulcerated and non-ulcerated foot. J Diabetes Complications. 2016 Sep-Oct;30(7):1293-9. doi: 10.1016/j.jdiacomp.2016.06.003. Epub 2016 Jun 8. PMID 27338509
- [Result] Chatzistergos PE, Naemi R, Chockalingam N. A method for subject-specific modelling and optimisation of the cushioning properties of insole materials used in diabetic footwear. Med Eng Phys. 2015 Jun;37(6):531-8. doi: 10.1016/j.medengphy.2015.03.009. Epub 2015 Apr 27. PMID 25937545
- [Result] Chatzistergos PE, Naemi R, Sundar L, Ramachandran A, Chockalingam N. The relationship between the mechanical properties of heel-pad and common clinical measures associated with foot ulcers in patients with diabetes. J Diabetes Complications. 2014 Jul-Aug;28(4):488-93. doi: 10.1016/j.jdiacomp.2014.03.011. Epub 2014 Mar 22. PMID 24795257
- [Result] Blazkiewicz M, Sundar L, Healy A, Ramachandran A, Chockalingam N, Naemi R. Assessment of lower leg muscle force distribution during isometric ankle dorsi and plantar flexion in patients with diabetes: a preliminary study. J Diabetes Complications. 2015 Mar;29(2):282-7. doi: 10.1016/j.jdiacomp.2014.10.007. Epub 2014 Oct 22. PMID 25454742
- [Result] Naemi, R., Linyard-Tough, K., Healy, A. and Chockalingam, N., 2015. The influence of slow recovery insole on plantar pressure and contact area during walking. Journal of Mechanics in Medicine and Biology, 15(02), p.1540005.
- See also: DiaBSmart — http://www.diabsmart.eu

RESULTS

PARTICIPANT FLOW:
Period: Six Months
Arm/Group | MCP Insole | PU Insole
Started | 41 | 41
Completed | 20 | 19
Not Completed | 21 | 22
Not completed — Did Not Show Up for Baseline Measurement | 7 | 6
Not completed — Lost to Follow-up | 14 | 16
Period: 12 Months
Arm/Group | MCP Insole | PU Insole
Started | 20 | 19
Completed | 16 | 14
Not Completed | 4 | 5
Not completed — Adverse Event | 2 | 2
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCP Insole | PU Insole | Total
Number analyzed (Participants) | 34 | 35 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 31 | 57
  >=65 years | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.7) | 56.1 (7.2) | 58.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 18 | 24 | 42
Height [Mean (Standard Deviation); unit: meters] | 1.63 (0.09) | 1.67 (0.08) | 1.65 (0.09)
Weight [Mean (Standard Deviation); unit: Kilogram] | 73 (11) | 77 (13) | 75 (12)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 13.3 (7.8) | 12.2 (6.0) | 12.8 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Postural Sway During Shod Standing
Description: Postural sway was recorded while standing on a pressure mat with eyes open for 30 seconds.
  Area of the center of pressure excursion
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | MCP Insole | PU Insole
Number analyzed (Participants) | 20 | 19
cm^2 | 4.3 (2.8) | 3.1 (2.7)

2. Secondary Outcome: Ankle Strength Left 1
Description: Strength during dorsi flexion using Citec Dynamometer
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: N
Arm/Group | MCP Insole | PU Insole
Number analyzed (Participants) | 20 | 19
N | 111 (40) | 116 (44)

3. Secondary Outcome: Ankle Strength Left 2
Description: Strength during plantar flexion using Citec Dynamometer
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: N
Arm/Group | MCP Insole | PU Insole
Number analyzed (Participants) | 20 | 19
N | 135 (47) | 140 (52)

4. Secondary Outcome: Ankle Strength Right 1
Description: Strength during dorsi flexion using Citec Dynamometer
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: N
Arm/Group | MCP Insole | PU Insole
Number analyzed (Participants) | 20 | 19
N | 107 (37) | 110 (39)

5. Secondary Outcome: Ankle Strength Right 2
Description: Strength during plantar flexion using Citec Dynamometer
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: N
Arm/Group | MCP Insole | PU Insole
Number analyzed (Participants) | 20 | 19
N | 132 (45) | 141 (47)

6. Other Pre Specified Outcome: Vibration Perception Threshold
Description: Average of left and right (8 measurement areas per foot)
Time Frame: Up to 6 months
Measure: Mean (Standard Deviation); unit: V
Arm/Group | MCP Insole | PU Insole
Number analyzed (Participants) | 20 | 19
V | 53 (19) | 65 (19)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | MCP Insole | PU Insole
All-Cause Mortality (participants affected / at risk) | 0/34 | 2/35
Serious Adverse Events (participants affected / at risk) | 2/34 | 2/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCP Insole (N=34) | PU Insole (N=35)
Ulceration (Skin and subcutaneous tissue disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Technical problems with in-shoe plantar pressure measurements lead to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes